CLINICAL TRIAL: NCT02786498
Title: A Blinded Exploratory Randomized Controlled Trial (RCT) to Determine Optimal Vitamin D3 Supplementation Strategies for Acute Fracture Healing
Brief Title: Optimal Vitamin D3 Supplementation Strategies for Acute Fracture Healing
Acronym: Vita-Shock
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Gerard Slobogean, Associate Professor of Orthopaedics, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: HP-00069705
Record Dates: First submitted 2016-05-11; First posted 2016-06-01 (Estimated); Results first posted 2021-04-01 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Fracture
Keywords: Tibial Shaft; Tibia; Femoral Shaft; Femur; Vitamin D; Fracture Healing
MeSH Terms: conditions — Fractures, Bone | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- High Loading Dose (Experimental): 150,000 IU loading dose vitamin D3 at enrolment and 6 weeks, plus daily dose placebo for 3 months.
  Interventions: Drug: Vitamin D3; Other: Placebo
- High Daily Dose (Experimental): Loading dose placebo at enrolment and 6 weeks, plus 4,000 IU vitamin D3 per day for 3 months.
  Interventions: Drug: Vitamin D3; Other: Placebo
- Low Daily Dose (Experimental): Loading dose placebo at enrolment and 6 weeks, plus 600 IU vitamin D3 per day for 3 months.
  Interventions: Drug: Vitamin D3; Other: Placebo
- Control Group (Placebo Comparator): Loading dose placebo at enrolment and 6 weeks, plus daily dose placebo for 3 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vitamin D3
  Arms: High Daily Dose; High Loading Dose; Low Daily Dose
Other: Placebo

SUMMARY:
The objective is to determine the effect of vitamin D3 supplementation on fracture healing at 3 months.

DETAILED DESCRIPTION:
Vitamin D supplements are increasingly being recommended to healthy adult fracture patients without an osteoporotic injury. Although this is a relatively new practice pattern, the basis for this adjunct therapy is grounded in the high hypovitaminosis D prevalence rates (up to 75%) among healthy adult fracture patients, and the strong biologic rationale for the role of vitamin D in fracture healing. Briefly, experimental animal studies have demonstrated that the concentration of vitamin D metabolites is higher at a fracture callus compared to the uninjured contralateral bone, vitamin D supplementation leads to decreased time to union and increased callus vascularity, and increases mechanical bone strength compared to controls. While evidence to confirm that vitamin D supplementation improves fracture healing in clinical studies does not exist, the pre-clinical data are compelling and worthy of further investigation.

With modern orthopaedic surgical care, rates of complications following tibia and femoral shaft fractures can be as high as 15%. Complications, including delayed union, nonunion, or infection often require secondary surgical procedures and result in profound personal and societal economic costs. While surgeons continue to seek advances in surgical technique, it is becoming increasingly obvious that innovations in orthopaedic techniques or implants are unlikely to eliminate complications. As a result, considerable attention is currently focused on adjunct biologic therapies, such as vitamin D.

A recent survey of 397 orthopaedic surgeons showed that only 26% routinely prescribe vitamin D supplementation to adult fracture patients. Of the 93 surgeons who indicated that they routinely prescribe vitamin D supplementation, 29 different dosing regimens were described ranging from low daily doses of 400 IU to loading doses of 600,000 IU. This suggests a high level of clinical uncertainty surrounding the use and optimal dose of vitamin D supplementation in adult fracture patients. If vitamin D supplementation improves fracture healing outcomes, then there is a large opportunity to increase its use; however, before widespread adoption occurs, research is needed to optimize the dosing strategy, establish the dosing safety in the immobilized fracture healing population, and overcome potential medication adherence issues among the often marginalized patients that suffer trauma.

The long-term goal of our research program is to conduct a large phase III RCT to determine which dose of vitamin D3 supplementation optimally improves acute fracture healing outcomes in healthy adult patients (18-50 years). The current proposed phase II exploratory trial will perform important preliminary work to test the central hypothesis that vitamin D3 dose and timing of administration is critical for improving fracture healing at 3 months. This trial will also inform the feasibility of the large phase III RCT.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men or women ages 18-50 years
2. Closed or low grade open (Gustilo type I or II) tibial or femoral shaft fracture
3. Fracture treated with a reamed, locked, intramedullary nail
4. Acute fracture (enrolled within 7 days of injury)
5. Provision of informed consent.

Exclusion Criteria:

1. Osteoporosis
2. Stress fractures
3. Elevated serum calcium (>10.5 mg/dL)
4. Atypical femur fractures as defined by American Society for Bone and Mineral Research (ASBMR) criteria
5. Pathological fractures secondary to neoplasm or other bone lesion
6. Patients with known or likely undiagnosed disorders of bone metabolism such as Paget's disease, osteomalacia, osteopetrosis, osteogenesis imperfecta etc.
7. Patients with hyperhomocysteinemia
8. Patients with an allergy to vitamin D or another contraindication to being prescribed vitamin D
9. Patients currently taking an over the counter multivitamin that contains vitamin D and are unable or unwilling to discontinue its use for this study
10. Patients who will likely have problems, in the judgment of the investigators, with maintaining follow-up
11. Pregnancy
12. Patients who are incarcerated
13. Patients who are not expected to survive their injuries
14. Other lower extremity injuries that prevent bilateral full weight-bearing by 6 weeks post-fracture.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Slobogean, MD, Principal Investigator — University of Maryland; Sheila Sprague, PhD, Principal Investigator — McMaster University
Locations (2):
- University of Maryland, R Adams Cowley Shock Trauma Center, Baltimore, Maryland, United States
- McMaster University, Center for Evidence-Based Orthopaedics, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Sprague S, Petrisor B, Scott T, Devji T, Phillips M, Spurr H, Bhandari M, Slobogean GP. What Is the Role of Vitamin D Supplementation in Acute Fracture Patients? A Systematic Review and Meta-Analysis of the Prevalence of Hypovitaminosis D and Supplementation Efficacy. J Orthop Trauma. 2016 Feb;30(2):53-63. doi: 10.1097/BOT.0000000000000455. PMID 26429406
- [Background] Omeroglu S, Erdogan D, Omeroglu H. Effects of single high-dose vitamin D3 on fracture healing. An ultrastructural study in healthy guinea pigs. Arch Orthop Trauma Surg. 1997;116(1-2):37-40. PMID 9006763
- [Background] Jingushi S, Iwaki A, Higuchi O, Azuma Y, Ohta T, Shida JI, Izumi T, Ikenoue T, Sugioka Y, Iwamoto Y. Serum 1alpha,25-dihydroxyvitamin D3 accumulates into the fracture callus during rat femoral fracture healing. Endocrinology. 1998 Apr;139(4):1467-73. doi: 10.1210/endo.139.4.5883. PMID 9528922
- [Background] Lidor C, Dekel S, Edelstein S. The metabolism of vitamin D3 during fracture healing in chicks. Endocrinology. 1987 Jan;120(1):389-93. doi: 10.1210/endo-120-1-389. PMID 3023034
- [Background] Lidor C, Dekel S, Hallel T, Edelstein S. Levels of active metabolites of vitamin D3 in the callus of fracture repair in chicks. J Bone Joint Surg Br. 1987 Jan;69(1):132-6. doi: 10.1302/0301-620X.69B1.3029136.
- [Background] Omeroglu H, Ates Y, Akkus O, Korkusuz F, Bicimoglu A, Akkas N. Biomechanical analysis of the effects of single high-dose vitamin D3 on fracture healing in a healthy rabbit model. Arch Orthop Trauma Surg. 1997;116(5):271-4. doi: 10.1007/BF00390051. PMID 9177802
- [Background] Study to Prospectively Evaluate Reamed Intramedullary Nails in Patients with Tibial Fractures Investigators; Bhandari M, Guyatt G, Tornetta P 3rd, Schemitsch EH, Swiontkowski M, Sanders D, Walter SD. Randomized trial of reamed and unreamed intramedullary nailing of tibial shaft fractures. J Bone Joint Surg Am. 2008 Dec;90(12):2567-78. doi: 10.2106/JBJS.G.01694. PMID 19047701
- [Background] Duan X, Al-Qwbani M, Zeng Y, Zhang W, Xiang Z. Intramedullary nailing for tibial shaft fractures in adults. Cochrane Database Syst Rev. 2012 Jan 18;1(1):CD008241. doi: 10.1002/14651858.CD008241.pub2. PMID 22258982
- [Background] Bhandari M, Guyatt GH, Tong D, Adili A, Shaughnessy SG. Reamed versus nonreamed intramedullary nailing of lower extremity long bone fractures: a systematic overview and meta-analysis. J Orthop Trauma. 2000 Jan;14(1):2-9. doi: 10.1097/00005131-200001000-00002. PMID 10630795
- [Background] Bonafede M, Espindle D, Bower AG. The direct and indirect costs of long bone fractures in a working age US population. J Med Econ. 2013;16(1):169-78. doi: 10.3111/13696998.2012.737391. Epub 2012 Oct 22. PMID 23035626
- [Background] Antonova E, Le TK, Burge R, Mershon J. Tibia shaft fractures: costly burden of nonunions. BMC Musculoskelet Disord. 2013 Jan 26;14:42. doi: 10.1186/1471-2474-14-42. PMID 23351958
- [Background] Kanakaris NK, Giannoudis PV. The health economics of the treatment of long-bone non-unions. Injury. 2007 May;38 Suppl 2:S77-84. doi: 10.1016/s0020-1383(07)80012-x. PMID 17920421
- [Background] Bhandari M, Schemitsch EH. Stimulation of fracture healing: osteobiologics, bone stimulators, and beyond. J Orthop Trauma. 2010 Mar;24 Suppl 1:S1. doi: 10.1097/BOT.0b013e3181d2d683. No abstract available. PMID 20182228
- [Background] Marsell R, Einhorn TA. Emerging bone healing therapies. J Orthop Trauma. 2010 Mar;24 Suppl 1:S4-8. doi: 10.1097/BOT.0b013e3181ca3fab. PMID 20182234
- [Background] Schoelles K, Snyder D, Kaczmarek J, Kuserk E, Erinoff E, Turkelson C, Coates V. The Role of Bone Growth Stimulating Devices and Orthobiologics in Healing Nonunion Fractures [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2005 Sep 21. Available from http://www.ncbi.nlm.nih.gov/books/NBK285118/ PMID 25879121
- [Background] Veitch SW, Findlay SC, Hamer AJ, Blumsohn A, Eastell R, Ingle BM. Changes in bone mass and bone turnover following tibial shaft fracture. Osteoporos Int. 2006;17(3):364-72. doi: 10.1007/s00198-005-2025-y. Epub 2005 Dec 15. PMID 16362144
- [Background] Hojsager FD, Rand MS, Pedersen SB, Nissen N, Jorgensen NR. Fracture-induced changes in biomarkers CTX, PINP, OC, and BAP-a systematic review. Osteoporos Int. 2019 Dec;30(12):2381-2389. doi: 10.1007/s00198-019-05132-1. Epub 2019 Aug 24. PMID 31446441
- [Derived] Sprague S, Bzovsky S, Connelly D, Thabane L, Adachi JD, Slobogean GP; Vita-Shock Investigators. Study protocol: design and rationale for an exploratory phase II randomized controlled trial to determine optimal vitamin D3 supplementation strategies for acute fracture healing. Pilot Feasibility Stud. 2019 Nov 22;5:135. doi: 10.1186/s40814-019-0524-4. eCollection 2019. PMID 31768262

RESULTS

PARTICIPANT FLOW:
Groups:
- High Loading Dose: 150,000 IU loading dose vitamin D3 at enrolment and 6 weeks, plus daily dose placebo for 3 months.
  Vitamin D3
  Placebo
- High Daily Dose: Loading dose placebo at enrolment and 6 weeks, plus 4,000 IU vitamin D3 per day for 3 months.
  Vitamin D3
  Placebo
- Low Daily Dose: Loading dose placebo at enrolment and 6 weeks, plus 600 IU vitamin D3 per day for 3 months.
  Vitamin D3
  Placebo
- Control Group: Loading dose placebo at enrolment and 6 weeks, plus daily dose placebo for 3 months.
  Placebo
Period: Overall Study
Arm/Group | High Loading Dose | High Daily Dose | Low Daily Dose | Control Group
Started | 27 | 24 | 24 | 27
Completed | 25 | 24 | 24 | 26
Not Completed | 2 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Loading Dose | High Daily Dose | Low Daily Dose | Control Group | Total
Number analyzed (Participants) | 27 | 24 | 24 | 27 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 24 | 24 | 27 | 102
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.4 (8.1) | 28.8 (7.3) | 31.1 (9.8) | 31.3 (7.9) | 29.65 (8.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 5 | 8 | 6 | 32
  Male | 14 | 19 | 16 | 21 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 0 | 1 | 5
  Not Hispanic or Latino | 25 | 22 | 24 | 26 | 97
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 11 | 11 | 10 | 15 | 47
  White | 14 | 11 | 13 | 10 | 48
  More than one race | 2 | 2 | 0 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 24 | 24 | 27 | 102
Smoking status [Count of Participants; unit: Participants]
  Current Smoker | 10 | 6 | 7 | 14 | 37
  Previous Smoker | 1 | 3 | 2 | 0 | 6
  Non-Smoker | 16 | 15 | 15 | 13 | 59
Fractured bone (Tibia) [Count of Participants; unit: Participants] | 11 | 9 | 10 | 11 | 41
Association for the Study of Internal fixation /Orthopaedic Trauma AssociationClassification (AO/OTA [Count of Participants; unit: Participants] — This system provides the clinician with standardized definitions so the verbal fracture description is precise and consistent from bone to bone and fracture to fracture. The system also provides a mechanism to convert the verbal description into an alphanumeric code to allow for data storage and future recall.
  The Numeric value indicates the bone while the values "A, B, C" indicate the type and severity of the fracture where A is a simple fracture and C is a complex fracture.
  Participants
    AO/OTA Class 32.A | 10 | 6 | 9 | 9 | 34
    AO/OTA Class 32.B | 4 | 4 | 5 | 3 | 16
    AO/OTA Class 32.C | 2 | 4 | 2 | 4 | 12
    AO/OTA Class 42.A | 7 | 3 | 3 | 6 | 19
    AO/OTA Class 42.B | 3 | 3 | 4 | 3 | 13
    AO/OTA Class 42.C | 1 | 4 | 1 | 2 | 8
Vitamin D3 deficient (25(OH)D Serum Levels ,20 ng/mL) [Count of Participants; unit: Participants] | 16 | 11 | 12 | 17 | 56

OUTCOME MEASURES:

1. Primary Outcome: Fracture Healing Will be Assessed Clinically Using Function IndeX for Trauma (FIX-IT)
Description: FIX-IT is a standardized measure of weight-bearing and pain in patients with lower extremity fractures, specifically tibia and femur fractures. The FIX-IT score ranges from 0 to 12 points in 2 domains: the ability to bear weight (maximum 6 points) and pain at the fracture site (maximum 6 points) The ability to bear weight is assessed through the single-leg stand and ambulation procedures. Pain is assessed through palpation and stress procedures. The scores in both domains, which are weighted equally, are summed to obtain the final total score; the maximum score of 12 indicates the highest level of function.
Time Frame: 3 months post-injury
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | High Loading Dose | High Daily Dose | Low Daily Dose | Control Group
Number analyzed (Participants) | 27 | 24 | 24 | 27
scores on a scale | 10.1 (2.5) | 9.7 (2.8) | 9.3 (3.3) | 9.0 (2.9)

2. Primary Outcome: Fracture Healing Will be Assessed Radiographically Using Radiographic Union Score for Tibial Fractures (RUST)
Description: Radiographic fracture healing was measured using the Radiographic Union Score for Tibial fractures (RUST), which assesses the presence of bridging callus or a persistent fracture line on each of four cortices. This method evaluates two orthogonal radiographic views; each cortex is attributed points ranging from 1 to 3. A fracture in the immediate postoperative period will receive the minimum score, 4, (1 point for each of the four cortices) and a fully consolidated or healed fracture will be assigned the maximum score, 12 (3 points on each of the four cortices).
Time Frame: 3 months post-injury
Measure: Mean (Standard Deviation); unit: Score on a scale 4-12
Arm/Group | High Loading Dose | High Daily Dose | Low Daily Dose | Control Group
Number analyzed (Participants) | 27 | 24 | 24 | 27
Score on a scale 4-12 | 11.0 (2.8) | 11.3 (2.9) | 11.0 (3.0) | 10.4 (2.5)

3. Primary Outcome: Fracture Healing Will be Assessed Biochemically Using Serum Levels of the Bone Turnover Marker (BTM) C-terminal Telopeptide of Type I Collagen (CTX)
Description: The BTM C-terminal telopeptide of type I collagen (CTX). CTX is a marker of bone resorption. Clinically important changes in the CTX markers are unknown; however, in a previous study of tibia fracture healing, Veitch et al observed concentrations of both bone turnover markers approximately 100% greater than baseline values.43 Given the large changes observed in these bone turnover markers, the same criteria will be applied for identifying a potentially clinically beneficial regimen and remain powered to detect a mean difference of 20% (SD 30%).
Time Frame: 3 months post-injury
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | High Loading Dose | High Daily Dose | Low Daily Dose | Control Group
Number analyzed (Participants) | 27 | 24 | 24 | 27
ng/mL | 0.59 (0.75) | 0.79 (0.93) | 0.67 (0.64) | 0.78 (0.97)

4. Primary Outcome: Fracture Healing Will be Assessed Biochemically Using Serum Levels of the Bone Turnover Marker N-terminal Propeptide of Type I Procollagen (P1NP)
Description: P1NP is a bone-formation marker and prior research has found that it is highest at 12 weeks after fractures of the tibial shaft and proximal femur.
Time Frame: 3 months post-injury
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | High Loading Dose | High Daily Dose | Low Daily Dose | Control Group
Number analyzed (Participants) | 27 | 24 | 24 | 27
ng/mL | 160.9 (140.1) | 187.8 (129.3) | 166.7 (115.8) | 140.7 (124.7)

5. Secondary Outcome: Serum Level of 25(OH)D
Description: Correlations will be assessed between participants' 25(OH)D levels at enrolment, changes in 25(OH)D levels from enrolment to 3 months, and 25(OH)D levels at 3 months and fracture healing
Time Frame: Up to 3 months post-injury
Population: Serum 25(OH)D Concentration by Treatment Group
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | High Loading Dose | High Daily Dose | Low Daily Dose | Control Group
Number analyzed (Participants) | 27 | 24 | 24 | 27
ng/mL
  Baseline | 18.8 (7.8) | 20.7 (9.6) | 19.7 (7.9) | 17.3 (7.5)
  Week 6 | 39.3 (17.8) | 38.4 (18.6) | 35.5 (22.5) | 26.1 (15.4)
  Month 3 | 39.9 (17.9) | 28.2 (20.7) | 38.1 (19.8) | 23.1 (19.0)

6. Secondary Outcome: Number of Participants With Adherence With Vitamin D Supplementation
Description: Will measure adherence with vitamin D supplementation based on participants self report at the 6 week and 3 month visits.
Time Frame: Up to 3 months post-injury
Measure: Count of Participants; unit: Participants
Arm/Group | High Loading Dose | High Daily Dose | Low Daily Dose | Control Group
Number analyzed (Participants) | 27 | 24 | 24 | 27
Participants
  6 Weeks | 19 | 20 | 18 | 22
  3 Months | 21 | 19 | 19 | 20

7. Secondary Outcome: Number of Participants With Adverse Events (AE)
Description: A count of the participants who experienced adverse events will measure participant safety
Time Frame: Up to 12 months post-injury
Measure: Count of Participants; unit: Participants
Arm/Group | High Loading Dose | High Daily Dose | Low Daily Dose | Control Group
Number analyzed (Participants) | 27 | 24 | 24 | 27
Participants | 9 | 10 | 11 | 14

8. Secondary Outcome: Serum Levels of Calcium
Description: Will measure participant safety
Time Frame: Up to 3 months post-injury
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | High Loading Dose | High Daily Dose | Low Daily Dose | Control Group
Number analyzed (Participants) | 27 | 24 | 24 | 27
mg/dL
  baseline | 9.1 (0.6) | 8.8 (0.7) | 8.3 (1.8) | 9.0 (0.6)
  Week 6 | 9.6 (0.3) | 9.6 (0.3) | 9.6 (0.4) | 9.6 (0.5)
  Month 3 | 9.5 (0.3) | 9.6 (0.5) | 9.7 (0.4) | 9.6 (0.3)

9. Secondary Outcome: Serum Levels of Parathyroid Hormone
Description: Helps the body to maintain stable levels of calcium in the blood
Time Frame: Up to 3 months post-injury
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | High Loading Dose | High Daily Dose | Low Daily Dose | Control Group
Number analyzed (Participants) | 27 | 24 | 24 | 27
pg/mL
  Baseline | 69.6 (39.0) | 64.7 (37.2) | 67.8 (35.1) | 60.3 (31.1)
  Week 6 | 41.9 (47.7) | 28.8 (32.2) | 68.0 (63.2) | 43.6 (47.7)
  Month 3 | 42.4 (39.6) | 71.0 (68.0) | 63.1 (48.1) | 74.6 (60.6)

10. Secondary Outcome: Count of Participants Who Completed Blood Measures
Description: Will measure participants adherence to the blood measures of the protocol.
Time Frame: Up to 3 months post-injury
Measure: Count of Participants; unit: Participants
Arm/Group | High Loading Dose | High Daily Dose | Low Daily Dose | Control Group
Number analyzed (Participants) | 27 | 24 | 24 | 27
Participants
  baseline | 26 | 24 | 24 | 26
  Week 6 | 21 | 20 | 15 | 22
  Month 3 | 19 | 11 | 17 | 15

11. Secondary Outcome: Count of Participants Who Completed Radiographic Imaging Measures
Description: Count of participants who completed radiographic imaging measures to determine participant protocol adherence and assists with identifying healing status
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | High Loading Dose | High Daily Dose | Low Daily Dose | Control Group
Number analyzed (Participants) | 27 | 24 | 24 | 27
Participants
  Baseline | 27 | 24 | 24 | 27
  Week 6 | 24 | 22 | 17 | 19
  Month 3 | 21 | 17 | 20 | 16
  Month 6 | 16 | 11 | 13 | 13
  Month 9 | 4 | 4 | 6 | 5
  Month 12 | 6 | 3 | 4 | 5

ADVERSE EVENTS:
Time Frame: 12 months after initial injury
Description: An Adverse Event (AE) is any symptom, sign, illness, or experience that develops or worsens in severity during the course of this study.
  AEs are classified as serious or non-serious.
Arm/Group | High Loading Dose | High Daily Dose | Low Daily Dose | Control Group
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/24 | 0/24 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/24 | 0/24 | 0/27
Other Adverse Events (participants affected / at risk) | 9/27 | 10/24 | 11/24 | 14/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Loading Dose (N=27) | High Daily Dose (N=24) | Low Daily Dose (N=24) | Control Group (N=27)
Fracture Healing Complication (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4) | 5 (5) | 6 (6) — fracture healing complications will be identified, and will include nonunion, delayed union, hardware failure 33 wound healing problems and infection (superficial and deep as defined by Centers for Disease Control and Prevention (CDC) criteria).
Non-study Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Vascular (Vascular disorders) | 2 (2) | 3 (3) | 0 (0) | 3 (3)
Gastrointestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Accident/Fall (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Recurrent Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retained Foreign Object (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Symptomatic Bullet
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sickle Cell Crisis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Re-operations for fracture healing complications (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) | 2 (2) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/98/NCT02786498/Prot_SAP_000.pdf